CLINICAL TRIAL: NCT03088943
Title: Assessment of Diastolic Function Using Intraoperative Transesophageal Echocardiography: Comparison of Mitral Annular Plane Velocity and Systolic Excursion Measured by Tissue Doppler Imaging vs. Speckle-Tracking
Brief Title: Intraoperative Diastolic Function by TDI and STE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick F Wouters, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Patrick F Wouters, MD PhD, Head of Anesthesiology, University Hospital, Ghent
Organization: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016/1550
Record Dates: First submitted 2017-02-14; First posted 2017-03-24 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2018-01

CONDITIONS: Echocardiography, Doppler; Echocardiography, Three-Dimensional; Echocardiography, Transesophageal; Echocardiography, Transthoracic

STUDY DESIGN:
Intervention Model Description: Patients will receive a series of perioperative echocardiographical measurements by TTE as well as TEE prior to induction, postinduction, and post cardiopulmonary bypass
Who Masked: Outcomes Assessor
Masking Description: Echo exams will be stored for later analysis by blinded assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TTE Apical 4 Chamber View (Other): Patients will receive TTE apical 4chamber echo examinations prior to induction and after induction
  Interventions: Other: TTE Apical 4 Chamber View
- TEE dTG View (Other): Patients will receive TEE deep transgastric echo examinations after induction and after cardiopulmonary bypass induction (paced at 80, 100, and 120 bpm)
  Interventions: Other: TEE dTG View
- TEE ME 4C View (Other): Patients will receive TEE midesophageal 4chamber echo examinations after induction and after cardiopulmonary bypass induction (paced at 80, 100, and 120 bpm)
  Interventions: Other: TEE ME 4C View

INTERVENTIONS:
Other: TTE Apical 4 Chamber View — We will measure a number of echocardiography parameters by TTE (apical 4 Chamber View) prior to and after induction
  Arms: TTE Apical 4 Chamber View
Other: TEE dTG View — We will measure a number of echocardiography parameters by TEE (dTG View) prior to cardiopulmonary bypass and after cardiopulmonary bypass (atrially paced at 80, 100, and 120 bpm)
  Arms: TEE dTG View
Other: TEE ME 4C View — We will measure a number of echocardiography parameters by TEE (ME 4C View) prior to cardiopulmonary bypass and after cardiopulmonary bypass (atrially paced at 80, 100, and 120 bpm)
  Arms: TEE ME 4C View

SUMMARY:
This project aims at exploring measures of diastolic function perioperatively.

DETAILED DESCRIPTION:
Perioperative echocardiographic quantification of myocardial function is of great importance in patient management and is increasingly being recommended intraoperatively in spite of some unresolved or under-explored issues. One such issue is the perioperative measurement of diastolic function. Diastolic dysfunction and diastolic heart failure - or as commonly referred to "heart failure with preserved ejection fraction (HFpEF)" - is responsible for some 35 to 50% of heart failures. Intraoperative measurements of diastolic function have a prognostic and management relevance for patients undergoing both cardiac and non-cardiac surgery. However, even recent guidelines on intraoperative transesophageal echocardiography (TEE) have neglected this topic, with the exception of the most recent, which briefly alluded to the role TEE can play in assessing diastolic function, but without addressing the issue of which measurements or views to use.

The clinically prevalent echocardiographic view for assessment of intraoperative diastolic function by tissue Doppler imaging (TDI) is the midesophageal 4-chamber (ME 4C) TEE view. This view, which looks at the heart from the left atrium, is the standard view for evaluating intraoperative global cardiac performance. However, the Doppler angle for assessing diastolic performance is generally much greater than 20° and, as Doppler techniques are known to be angle dependent based on the Doppler equation, using this view may relevantly underestimate TDI velocities. Views from the apex of the heart (i.e. both the deep transgastric long axis view [dTG LAX] TEE view as well as the apical 4-chamber [AP 4C] transthoracic echocardiography (TTE) view) have a cosine angle towards the mitral annular plane excursion near zero, thereby allowing valid measurements according to the Doppler equation. However, TDI velocities are often - and potentially erroneously - reported from the ME 4C TEE view.

The objective of this project is to address a number of important clinical topics regarding diastolic dysfunction in TEE.

Two main objectives will be examined:

* Assess whether or not tissue doppler imaging (TDI) measurements of mitral annular plane velocities and systolic excursion in the midesophageal 4-chamber TEE view (ME 4C) significantly underestimate diastolic cardiac performance compared to the deep transgastric long axis TEE view (dTG LAX) due to intrinsic misalignment of the doppler beam.

  [i.e. is there a technological limitation?]
* Assess whether or not the difference in mitral annular plane velocities and systolic excursion between the ME 4C and dTG LAX will be underestimated using TDI compared to values derived from speckle tracking echocardiography (STE).

  [i.e. if there is a technological limitation, does STE show more consistency?]

Two secondary objectives will be examined:

* Determine the influence of frame rates (temporospatial resolution) on STE-derived mitral annular velocities and systolic excursion by conducting STE measurement post cardiopulmonary Bypass (CPB) in atrially paced patients in the 1. midesophageal 4 chamber view (ME 4C) and 2. deep transgastric long axis view (dTG LAX).

  [i.e. if ST shows more consistency, what are its limitations?]
* Confirm the existence of and explore potential reasons (anesthesia, ventilation, TTE vs. TEE, Doppler alignment) for differences in mitral annular plane velocities and systolic excursion observed preoperatively (i.e. by cardiologists) and intraoperatively (i.e. by anesthetists, intensivists). Specifically, we will compare these values in four views: 1. apical 4-chamber view in TTE (AP 4C) preinduction, 2. apical 4-chamber view in TTE (AP 4C) postinduction, 3. midesophageal 4 chamber view (ME 4C) postinduction, and 4. Deep transgastric long axis view (dTG LAX) postinduction.

  [i.e. what is the relative contribution of the ignoring the misalignment in angulation compared to other intraoperative factors in explaining the observed underestimation of diastolic velocities and distances seen by cardiologists (AP 4C TTE view) and anesthetist's/intensivist's (ME 4C TEE view)?]

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* undergoing cardiac surgery, and
* routinely receiving TEE for the surgical procedure, independent of the study.

Exclusion Criteria:

* atrial flutter or fibrillation
* severe mitral calcification
* cancelled surgery
* unwilling or unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
mean early diastolic mitral annular plane velocity (E') | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  (E'lateral + E'medial)/2; by TDI and STE

SECONDARY OUTCOMES:
mean late (atrial) diastolic mitral annular plane velocity (A') | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  (A'lateral + A'medial)/2; by TDI and STE
mean early diastolic mitral annular plane velocity/mean late (atrial) diastolic mitral annular plane velocity (E'/A') | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  [(E'lateral + E'medial)/2] / [(A'lateral + A'medial)/2]; by TDI and STE
mean early diastolic mitral inflow velocity/mean early diastolic mitral annular plane velocities; (E/E') | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  E/[(E'lateral + E'medial)/2]; by doppler, TDI, and STE
Peak systolic mitral annular velocity (S') | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  by TDI and STE
Displacement by Mitral Annular Plane Systolic Excursion (MAPSE) | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  (MAPSEmedial + MAPSElateral)/2
Displacement by Tricuspid Annular Place Systolic Excursion (TAPSE) | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  only laterally
Displacement of Mitral Annular Plane (by speckle-tracking software) | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  using tissue Motion annular displacement (TMAD) in Cardiovascular Ultrasound Quantification Software (QLAB)
Displacement of Tricuspid Annular Plane (by speckle-tracking software) | immediately during echo exam while in the operating room; i.e. preinduction (TTE AP 4C), postinduction (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view), post-CPB (TTE AP 4C view, TEE ME 4C view, TEE dTG LAX view)
  using tissue Motion annular displacement (TMAD) in Cardiovascular Ultrasound Quantification Software (QLAB)
3D volumes of left ventricle | immediately during echo exam while in the operating room; i.e. postinduction (TEE ME 4C view), post-CPB (TEE ME 4C view)
  using 4-beat ECG-gated image acquisition
3D volumes of right ventricle | immediately during echo exam while in the operating room; i.e. postinduction (TEE ME 4C view), post-CPB (TEE ME 4C view)
  using 4-beat ECG-gated image acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F Wouters, MD, PhD, Study Director — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, East-Flanderse, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Mauermann E, Bouchez S, Bove T, Vandenheuvel M, Wouters P. Assessing Left Ventricular Early Diastolic Velocities With Tissue Doppler and Speckle Tracking by Transesophageal and Transthoracic Echocardiography. Anesth Analg. 2021 May 1;132(5):1400-1409. doi: 10.1213/ANE.0000000000005469. PMID 33857980